CLINICAL TRIAL: NCT05273190
Title: Vibrotactile Stimulation of the Larynx to Treat Unexplained Chronic Cough
Brief Title: Stimulation of the Larynx to Treat Unexplained Chronic Cough
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT-2020-28903; R34HL174877 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-03-10 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cough
Keywords: Chronic cough
MeSH Terms: conditions — Cough; Chronic Cough

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Vibrotactile Stimulation (Experimental)
  Interventions: Device: Vibrotactile Stimulation

INTERVENTIONS:
Device: Vibrotactile Stimulation — Small electric motors, similar to a vibrating cell phone or gaming joystick, deliver vibration to the throat. Participants will assess cough symptoms throughout the study period.

SUMMARY:
Researchers will test the effect of non-invasive vibrotactile stimulation of the larynx on symptom severity of unexplained chronic cough.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-88
* >8 weeks of cough
* Cough visual analogue scale (VAS): Rating of 30 or greater on a 0-100 cough severity scale
* Ability to provide informed consent and independently complete questionnaires
* Ability to read and speak English

Exclusion Criteria:

* Electronic implants (e.g., pacemaker)
* Currently doing speech therapy for cough
* Contraindications to safe or effective VTS device use
* No regular access to wifi internet Neuromuscular impairment that may affect cough/laryngeal sensation and/or function (e.g., multiple system atrophy, Parkinson, CVA, vocal fold paralysis or paresis)
* Untreated carotid disease
* BMI > 40 (for transmission of VTS through soft tissue)
* Current or recent (quit < 3 months ago) smoking
* Known currently infectious cause for cough (e.g., TB, pertussis, COVID)
* History of known or suspected aspiration pneumonia
* Diagnosis or clinical suspicion of chronic obstructive pulmonary disease (COPD)
* Diagnosis or clinical suspicion of interstitial lung disease (ILD)
* Unmanaged reflux
* Unmanaged allergies/postnasal drip

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess usability of VTS device | 3-7 weeks
  % of participants indicating agree or strongly agree with statements of usability
Impact of VTS on cough symptoms | 3-7 weeks
  Pre-post comparison of LCQ scores

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Misono, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States